CLINICAL TRIAL: NCT00552058
Title: Phase IIIb, Multinational, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of Certolizumab Pegol, a Pegylated Fab' Fragment of a Humanized Anti-Tumor Necrosis Factor(TNF)-Alpha Monoclonal Antibody, Administered in Subjects With Moderately to Severely Active Crohn's Disease.
Brief Title: Study to Evaluate Efficacy and Safety of Certolizumab Pegol for Induction of Remission in Patients With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C87085; 2007-001913-41 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2007-10-18; First posted 2007-11-01 (Estimated); Results first posted 2010-12-30 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2011-10

CONDITIONS: Crohn Disease
Keywords: CDP 870; Certolizumab Pegol; CIMZIA ®; Crohn's disease; Induction; Clinical remission; Clinical response
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab pegol (Experimental): Certolizumab pegol 400 mg for subcutaneous (sc) injection
  Interventions: Biological: certolizumab pegol (CDP870, CZP)
- Placebo (Placebo Comparator): Placebo, saline solution for sc injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: certolizumab pegol (CDP870, CZP) — Certolizumab Pegol 400 mg CZP sc injection 2 x 1 mL CZP (200 mg/mL) at Week 0, 2, and 4
  Other Names: CIMZIA ®; CDP870; CZP
  Arms: Certolizumab pegol
Other: Placebo — Saline 0.9% sc injection 2 x 1 mL Placebo at Week 0, 2 and 4
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate efficacy of certolizumab pegol in inducing clinical remission in patients with moderate to severe Crohn's disease as compared with placebo based on Crohn's Disease Activity Index (CDAI) score at Week 6.

ELIGIBILITY:
Inclusion Criteria:

* male/female
* 18 - 75 years inclusive
* diagnosis of Crohn's disease confirmed
* moderate to severe disease activity (Crohn's Disease Activity Index (CDAI) 225 - 450)
* no previous treatment with anti-tumor necrosis factor (anti-TNF) medications

Exclusion Criteria:

* previous participation in a certolizumab pegol study
* general exclusion criteria as common for studies in this indication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (116):
- United States (24):
  - Pell City, Alabama
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Hollywood, Florida
  - Jacksonville, Florida
  - New Port Richey, Florida
  - Winter Park, Florida
  - Chicago, Illinois
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Monroe, Louisiana
  - Annapolis, Maryland
  - Towson, Maryland
  - Chesterfield, Michigan
  - West Bloomfield, Michigan
  - Rochester, Minnesota
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Lancaster, Pennsylvania
  - Germantown, Tennessee
  - Norfolk, Virginia
  - Seattle, Washington
- Australia (10):
  - Concord, New South Wales
  - Box Hill, Victoria
  - Footscray, Victoria
  - Parkville, Victoria
  - Adelaide
  - Bankstown
  - Clayton
  - Fitzroy
  - Fremantle
  - Garran
- Vienna, Austria
- Belgium (6):
  - Bonheiden
  - Brussels
  - Ghent
  - Leuven
  - Liège
  - Roeselare
- Brazil (8):
  - Belo Horizonte, Minas Gerais
  - Curitiba
  - Goiânia
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
  - Santos
  - São Paulo
- Canada (8):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Calgary
- Chile (2):
  - Santiago
  - Viña del Mar
- Czechia (5):
  - Hradec Králové
  - Hradek Kralove
  - Prague
  - Ústí nad Orlicí
  - Zlín
- Estonia (2):
  - Tallinn
  - Tartu
- Mikkeli, Finland
- Germany (9):
  - Berlin
  - Frankfurt
  - Freiburg im Breisgau
  - Homburg
  - Jena
  - Kiel
  - München
  - Ulm
  - Wilhelmshaven
- Hungary (5):
  - Budapest
  - Győr
  - Nagykanizsa
  - Szeged
  - Szombathely
- Israel (9):
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petha Tikva
  - Rehovot
  - Tel Aviv
  - Ẕerifin
- Italy (3):
  - Bologna
  - Padua
  - Roma
- Latvia (2):
  - Riga
  - Valmiera
- New Zealand (5):
  - Milford, Auckland
  - Newton, Wellington Region
  - Auckland
  - Christchurch
  - Hamilton
- Poland (4):
  - Częstochowa
  - Lodz
  - Warsaw
  - Wroclaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Constanța
- Russia (3):
  - Kazan'
  - Moscow
  - Saint Petersburg
- Ukraine (6):
  - Dniepropetrovsk
  - Donetsk
  - Kiev
  - Kyiv
  - Lviv
  - Simferopol

REFERENCES:
- [Result] Sandborn WJ, Schreiber S, Feagan BG, Rutgeerts P, Younes ZH, Bloomfield R, Coteur G, Guzman JP, D'Haens GR. Certolizumab pegol for active Crohn's disease: a placebo-controlled, randomized trial. Clin Gastroenterol Hepatol. 2011 Aug;9(8):670-678.e3. doi: 10.1016/j.cgh.2011.04.031. Epub 2011 May 13. PMID 21642014
- [Derived] Sandborn WJ, Melmed GY, McGovern DP, Loftus EV Jr, Choi JM, Cho JH, Abraham B, Gutierrez A, Lichtenstein G, Lee SD, Randall CW, Schwartz DA, Regueiro M, Siegel CA, Spearman M, Kosutic G, Pierre-Louis B, Coarse J, Schreiber S. Clinical and demographic characteristics predictive of treatment outcomes for certolizumab pegol in moderate to severe Crohn's disease: analyses from the 7-year PRECiSE 3 study. Aliment Pharmacol Ther. 2015 Aug;42(3):330-42. doi: 10.1111/apt.13251. Epub 2015 Jun 1. PMID 26031921
- [Derived] Sandborn WJ, Lee SD, Randall C, Gutierrez A, Schwartz DA, Ambarkhane S, Kayhan C, Pierre-Louis B, Schreiber S, Lichtenstein GR. Long-term safety and efficacy of certolizumab pegol in the treatment of Crohn's disease: 7-year results from the PRECiSE 3 study. Aliment Pharmacol Ther. 2014 Oct;40(8):903-16. doi: 10.1111/apt.12930. Epub 2014 Aug 22. PMID 25146586
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants flow shows all subjects randomized. Safety analyses are based on actual treatment received; 1 subject randomized to placebo did not receive any treatment thus would be excluded due to the definition of the safety population.
Period: Overall Study
Arm/Group | Certolizumab Pegol | Placebo
Started | 223 | 216
Completed | 207 | 192
Not Completed | 16 | 24
Not completed — Adverse Event | 8 | 7
Not completed — Lack of Efficacy | 1 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Other: Protocol Violation | 0 | 1
Not completed — Other: Non Compliance | 1 | 2
Not completed — Other: Crossed Over to a Follow-up Study | 0 | 1
Not completed — Other: Low CDAI score, entry violation | 0 | 1
Not completed — Other: Positive Stool Result | 0 | 1
Not completed — Other: Randomized in error | 0 | 1
Not completed — Other: Sponsors Decision | 0 | 1
Not completed — Other: Early Roll Over | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Certolizumab Pegol | Placebo | Total
Number analyzed (Participants) | 223 | 215 | 438
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 213 | 205 | 418
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (12.63) | 38.8 (12.76) | 37.5 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 125 | 243
  Male | 105 | 90 | 195
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 83
  Estonia | 2 | 2 | 4
  Ukraine | 10 | 13 | 23
  Austria | 5 | 3 | 8
  Russian Federation | 8 | 7 | 15
  Israel | 12 | 10 | 22
  Italy | 5 | 8 | 13
  Czech Republic | 13 | 9 | 22
  Hungary | 25 | 25 | 50
  Canada | 34 | 32 | 66
  Poland | 15 | 15 | 30
  Belgium | 7 | 7 | 14
  Brazil | 16 | 10 | 26
  Romania | 4 | 3 | 7
  Australia | 8 | 12 | 20
  Latvia | 3 | 5 | 8
  Germany | 4 | 4 | 8
  New Zealand | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in Clinical Remission at Week 6
Description: The percentage of subjects in clinical remission at Week 6 (clinical remission is defined as a total Crohn's Disease Activity Index (CDAI) score of 150 points or less). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 6
Population: Of the 223 (Certolizumab Pegol 400 mg) and 216 (Placebo) subjects randomized, 215 and 209 subjects are included in the Intent-to-treat (ITT) population, respectively. ITT population: subjects who received at least one dose of study drug, and who had at least one efficacy measurement after first dose.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 31.6 [25.4 to 37.8] | 25.4 [19.5 to 31.3]

2. Secondary Outcome: Percentage of Subjects Achieving a Clinical Response at Week 6
Description: The percentage of subjects achieving a clinical response at Week 6 (clinical response is defined as at least a 100-point decrease from the Week 0 Crohn's Disease Activity Index (CDAI) score). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0, Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 40.5 [33.9 to 47.0] | 34.0 [27.6 to 40.4]

3. Secondary Outcome: Percentage of Subjects in Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week 6
Description: The percentage of subjects in Inflammatory Bowel Disease Questionnaire (IBDQ) remission at Week 6 (IBDQ remission is defined as a total IBDQ score of 170 points or more). The IBDQ Global Score is the sum of 32 responses, each ranging from 0 to 7, thus the Global Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 36.7 [30.3 to 43.2] | 28.7 [22.6 to 34.8]

4. Secondary Outcome: Change in Total Crohn's Disease Activity Index (CDAI) Score From Week 0 to Week 6
Description: The change in total Crohn's Disease Activity Index (CDAI) score from Week 0 to Week 6. CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0 to Week 6
Population: Of the 215 (Certolizumab Pegol 400 mg) and 209 (Placebo) subjects in the Intent-to-treat (ITT) population, 192 and 183 subjects respectively are included in this summary and have assessments at both Weeks 0 and 6. ITT population: subjects who received at least one dose of study drug, and who had at least one efficacy measurement after first dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 192 | 183
score on a scale | -96.7 (100.86) | -73.1 (95.07)

5. Secondary Outcome: Change in Harvey Bradshaw Index (HBI) Score From Week 0 to Week 6
Description: The change in Harvey Bradshaw Index (HBI) score from Week 0 to Week 6. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (score 1 per item). The first three items are scored for the previous day. Lower scores indicated better well being.
Time Frame: Week 0 to Week 6
Population: Of the 215 (Certolizumab Pegol 400 mg) and 209 (Placebo) subjects in the Intent-to-treat (ITT) population, 196 and 187 subjects respectively are included in this summary and have assessments at both Weeks 0 and 6. ITT population: subjects who received at least one dose of study drug, and who had at least one efficacy measurement after first dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 196 | 187
score on a scale | -3.3 (4.00) | -2.6 (3.90)

6. Secondary Outcome: Percentage of Subjects in Clinical Remission at Week 2
Description: The percentage of subjects in clinical remission at Week 2 (clinical remission is defined as a total Crohn's Disease Activity Index (CDAI) score of 150 points or less). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 23.3 [17.6 to 28.9] | 15.8 [10.8 to 20.7]

7. Secondary Outcome: Percentage of Subjects in Clinical Remission at Week 4
Description: The percentage of subjects in clinical remission at Week 4 (clinical remission is defined as a total Crohn's Disease Activity Index (CDAI) score of 150 points or less). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 26.5 [20.6 to 32.4] | 19.1 [13.8 to 24.5]

8. Secondary Outcome: Percentage of Subjects Achieving a Clinical Response at Week 2
Description: The percentage of subjects achieving a clinical response at Week 2 (clinical response is defined as at least a 100-point decrease from the Week 0 Crohn's Disease Activity Index (CDAI) score). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0, Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 33.0 [26.7 to 39.3] | 20.1 [14.7 to 25.5]

9. Secondary Outcome: Percentage of Subjects Achieving a Clinical Response at Week 4
Description: The percentage of subjects achieving a clinical response at Week 4 (clinical response is defined as at least a 100-point decrease from the Week 0 Crohn's Disease Activity Index (CDAI) score). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0, Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 35.3 [29.0 to 41.7] | 26.3 [20.3 to 32.3]

10. Secondary Outcome: Change in Total Crohn's Disease Activity Index (CDAI) Score From Week 0 to Week 2
Description: The change in total Crohn's Disease Activity Index (CDAI) score from Week 0 to Week 2. CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0 to Week 2
Population: Of the 215 (Certolizumab Pegol 400 mg) and 209 (Placebo) subjects in the Intent-to-treat (ITT) population, 204 and 198 subjects respectively are included in this summary and have assessments at both Weeks 0 and 2. ITT population: subjects who received at least one dose of study drug, and who had at least one efficacy measurement after first dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 204 | 198
score on a scale | -72.6 (81.26) | -41.8 (82.06)

11. Secondary Outcome: Change in Total Crohn's Disease Activity Index (CDAI) Score From Week 0 to Week 4
Description: The change in total Crohn's Disease Activity Index (CDAI) score from Week 0 to Week 4. CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0, Week 4
Population: Of the 215 (Certolizumab Pegol 400 mg) and 209 (Placebo) subjects in the Intent-to-treat (ITT) population, 198 and 184 subjects respectively are included in this summary and have assessments at both Weeks 0 and 4. ITT population: subjects who received at least one dose of study drug, and who had at least one efficacy measurement after first dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 198 | 184
score on a scale | -88.8 (91.36) | -65.7 (83.06)

12. Secondary Outcome: Percentage of Subjects in Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week 2
Description: The percentage of subjects in Inflammatory Bowel Disease Questionnaire (IBDQ) remission at Week 2 (IBDQ remission is defined as a total IBDQ score of 170 points or more). The IBDQ Global Score is the sum of 32 responses, each ranging from 0 to 7, thus the Global Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 25.6 [19.7 to 31.4] | 18.2 [13.0 to 23.4]

13. Secondary Outcome: Percentage of Subjects in Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week 4
Description: The percentage of subjects in Inflammatory Bowel Disease Questionnaire (IBDQ) remission at Week 4 (IBDQ remission is defined as a total IBDQ score of 170 points or more). The IBDQ Global Score is the sum of 32 responses, each ranging from 0 to 7, thus the Global Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 215 | 209
percentage of subjects | 33.5 [27.2 to 39.8] | 23.9 [18.1 to 29.7]

14. Secondary Outcome: Percentage of Subjects in Subgroup With Less Than 10 mg/L C-reactive Protein (CRP) at Entry Who Are in Clinical Remission at Week 6
Description: The percentage of subjects in the subgroup with less than 10 mg/L of C-reactive Protein (CRP) at Entry who are in clinical remission at Week 6 (clinical remission is defined as a total Crohn's Disease Activity Index (CDAI) score of 150 points or less). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 6
Population: Of 215 (Certolizumab Pegol 400 mg) and 209 (Placebo) subjects in the Intent-to-treat (ITT) population, 122 and 113 subjects are in the less than 10 mg/L C-reactive Protein (CRP) subgroup at Entry, respectively. ITT population: subjects who received at least one dose of study drug, and who had at least one efficacy measurement after first dose.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 122 | 113
percentage of subjects | 30.3 [22.2 to 38.5] | 30.1 [21.6 to 38.5]

15. Secondary Outcome: Percentage of Subjects in Subgroup With 10 mg/L or Greater C-reactive Protein (CRP) at Entry Who Are in Clinical Remission at Week 6
Description: The percentage of subjects in the subgroup with 10 mg/L or greater C-reactive Protein (CRP) at Entry in clinical remission at Week 6 (clinical remission is defined as a total Crohn's Disease Activity Index (CDAI) score of 150 points or less). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 6
Population: Of the 215 (Certolizumab Pegol 400 mg) and 209 (Placebo) subjects in the Intent-to-treat (ITT) population, 93 and 96 subjects are in the 10 mg/L or greater C-reactive Protein (CRP) subgroup at Entry, respectively. ITT population: subjects who received at least one dose of study drug, and who had at least one efficacy measurement after first dose.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 93 | 96
percentage of subjects | 33.3 [23.8 to 42.9] | 19.8 [11.8 to 27.8]

16. Secondary Outcome: Percentage of Subjects in Subgroup With Less Than 10 mg/L C-reactive Protein (CRP) at Entry Achieving a Clinical Response at Week 6
Description: The percentage of subjects in the subgroup with less than 10 mg/L C-reactive Protein (CRP) at Entry achieving a clinical response at Week 6 (clinical response is defined as at least a 100-point decrease from the Week 0 Crohn's Disease Activity Index (CDAI) score). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0, Week 6
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 122 | 113
percentage of subjects | 37.7 [29.1 to 46.3] | 35.4 [26.6 to 44.2]

17. Secondary Outcome: Percentage of Subjects in Subgroup With 10 mg/L or Greater C-reactive Protein (CRP) at Entry Achieving a Clinical Response at Week 6
Description: The percentage of subjects in the subgroup with 10 mg/L or greater C-reactive Protein (CRP) at Entry achieving a clinical response at Week 6 (clinical response is defined as at least a 100-point decrease from the Week 0 Crohn's Disease Activity Index (CDAI) score). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 points or below indicates clinical remission and a score above 450 points indicates extremely severe disease.
Time Frame: Week 0, Week 6
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol | Placebo
Number analyzed (Participants) | 93 | 96
percentage of subjects | 44.1 [34.0 to 54.2] | 32.3 [22.9 to 41.6]

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Arm/Group | Certolizumab Pegol | Placebo
Serious Adverse Events (participants affected / at risk) | 12/223 | 8/215
Other Adverse Events (participants affected / at risk) | 48/223 | 42/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=223) | Placebo (N=215)
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 3 (3) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (4) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 2 (2) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
HIV INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PERIANAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FISTULA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=223) | Placebo (N=215)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (10) | 8 (8)
NAUSEA (Gastrointestinal disorders) | 9 (9) | 10 (11)
FATIGUE (General disorders) | 9 (9) | 2 (2)
PYREXIA (General disorders) | 7 (9) | 10 (14)
URINARY TRACT INFECTION (Infections and infestations) | 7 (7) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6)
HEADACHE (Nervous system disorders) | 12 (13) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.